CLINICAL TRIAL: NCT02934204
Title: Temozolomide in Treatment of Patients With Primary Central Nervous System Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDREC2015431H(R1)
Record Dates: First submitted 2016-10-13; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-05

CONDITIONS: Primary CNS Lymphoma
Keywords: PCNSL; DLBCL; methotrexate; temozolomide
MeSH Terms: interventions — Methotrexate; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MTX and Temozolomide (Experimental): Induction therapy:
  Methotrexate 3.5g/m2 ivgtt d1 2weeks/cycle，total 8 cycles Temozolomide 150mg/m2 po d1-5 4weeks/cycle, total 4 cycles
  Consolidation therapy:
  PCNSL patients achieve CR,Temozolomide 150mg/m2 po d1-5 4weeks/cycle, total 12 cycles
  Interventions: Drug: methotrexate; Drug: temozolomide

INTERVENTIONS:
Drug: methotrexate
Drug: temozolomide

SUMMARY:
Consolidation treatment for Primary Central Nervous System Diffuse Large B cell Lymphoma(PCNSL)patients remains to be defined.Here we designed a tolerated treatment of HDMTX plus Temozolomide,followed by consolidation with Temozolomide in PCNSL patients.

ELIGIBILITY:
Inclusion Criteria:

- (1) histology confirmed to be PCNSL. (2) lymphoma invasion in brain, meninges, cerebrospinal fluid, eye organ. (3) ECOG score less than 3 points (4) at least 1 of the lesions can be evaluated with a double diameter. (5) the life expectancy of more than 6 months. (6) less or equal to 75 years,or more or equal to 18 years. (7) to be able to comply with the requirements of the study and follow-up procedures.

(8) to sign the consent form to participate in the study. (9) having adequate organ function, defined as follows: Liver function, serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) equal to or less than 2 times the upper limit of normal (ULN).

Bone marrow function: absolute neutrophil count more or equal to 1500/L, platelet count more than 100000/L,hemoglobin was greater than 9 g/dL.

Renal function, serum creatinine or creatinine clearance rate (less than 1.5ULN Cockcroft-Gault formula based on the improvement of more than 50ml/min).

(10) women with childbearing potential must start to get the test results of serum / urine pregnancy test negative within 48 hours prior to study. Postmenopausal women who have at least 12 months of menopause can be treated as non fertile.

Exclusion Criteria:

* (1) patients with a history of other malignancies within five years (except for the full treatment of cervical carcinoma in situ or basal cell carcinoma or squamous cell skin cancer).

  (2) had previously been treated with total cranial irradiation. (3) the upper digestive tract is lack of physical integrity, or suffering from malabsorption syndrome, or oral drug, or active gastric ulcer.

  (4) suffering from any unstable systemic diseases (including active infection, significant cardiovascular disease, any significant liver and kidney or metabolic disorders), metabolic disorders, physical examination results or laboratory examination results of contraindication to the use of drugs, or may affect the treatment results of interpretation or increase the risk of complications in treatment of risk (5) patients with human immunodeficiency virus (HIV) transmitted in the form of blood or other body fluids.

  (6) women in pregnancy and lactation. (7) women of childbearing age who do not want to use contraceptive measures during the study period and have sexual capacity of men.

  (8) patients who do not want to sign informed consent. (9) patients who were not willing to follow up. (10) for any drugs or excipients of allergy. Exit the case: no matter what reason patients withdrew from the study of cases in time will be postponed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
event free survival | 3 year

SECONDARY OUTCOMES:
Chronic neurotoxicity | 3 year
Overall survival | 3 year
Completed response | 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong general hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No